CLINICAL TRIAL: NCT01012999
Title: Pain Control and Patient Satisfaction: a Dosing Study to Determine a Safe and Effective Dose of Intra-nasal Sufentanil to Treat Emergency Department Patients With Moderate to Severe Pain Due to Extremity Trauma
Brief Title: A Dosing and Efficacy Study of Intra-nasal Sufentanil for Moderate to Severe Pain
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Robert Stephen, MD, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32225
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Pain; Opiate
Keywords: acute pain, intranasal, sufentanil,; Acute pain control with an intranasal opiate
MeSH Terms: conditions — Pain; Acute Pain | interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intranasal sufentanil, pain relief (Experimental): Intranasal sufentanil administered at a dose of 0.5 mcg/kg times one dose at beginning of thirty minute period
  Interventions: Drug: sufentanil

INTERVENTIONS:
Drug: sufentanil — Intra-nasal delivery, dosing range 0.5 mcg/kg, administered once at the beginning of the 30 minute study period
  Other Names: Sufenta

SUMMARY:
The purpose of this study is to determine the appropriate dose and effectiveness of intra-nasal administration of a potent narcotic, sufentanil, for the treatment of moderate to severe pain due to broken bone(s) in the arm or leg.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older;
* isolated traumatic injury to upper or lower extremity;
* alert and oriented to name, date, place; patient has a numeric pain score of 5 or higher;
* speaks English as their primary language;
* female patients are on birth control, menopausal, or are sterile (hysterectomy, tubal ligation)

Exclusion Criteria:

* injury isolated to a finger or toe;
* previous nasal or sinus surgery; chronic nasal problem;
* acute nasal problem (ie epistaxis, upper respiratory infection, sinusitis);
* pregnant; prisoner; allergy to sufentanil, fentanyl, or alfentanil; history of analgesic abuse or dependency;
* presence of other painful injuries; systolic Blood Pressure less than 100 mm Hg;
* patient seems or is confused or has a head injury; room air oxygenation less than 95%;
* patient has chronic obstructive pulmonary disease, severe asthma, oxygen-dependent pulmonary disease;
* impaired hepatic or renal function (obtained clinically or by history);
* weight more than 230 lbs (100 kg);
* alcohol or drug intoxication (per patient admission or clinical assessment of physician);
* elderly (> 70 years)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stephen, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Over a 2 year period we recruited 16 patients who presented to a single Emergency Department.
Groups:
- Intranasal Sufentanil, Pain Relief: Patients with a suspected acute bony injury to an extremity and in moderate to severe pain.
  Intranasal administration, 0.5 mcg/kg, one time dose.
Period: Overall Study
Arm/Group | Intranasal Sufentanil, Pain Relief
Started | 16
Completed | 15
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Patients with a suspected acute bony injury to an extremity and in moderate to severe pain.
  Intranasal administration, 0.5-0.9 mcg/kg, maximum dosage of 100 mcg
Groups:
- Intranasal Sufentanil, Pain Relief: Patients with a suspected acute bony injury to an extremity and in moderate to severe pain.
  Intranasal administration, 0.5 mcg/kg to an extremity and in moderate to severe pain, one time dose.
Arm/Group | Intranasal Sufentanil, Pain Relief
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at Thirty Minutes
Description: Measured pain relief on a visual analog scale (0-10- ten being the worst pain and zero being no pain at all).
Time Frame: 30 min post dose
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Intranasal Sufentanil, Pain Relief: Patients with a suspected acute bony injury to an extremity and in moderate to severe pain
Arm/Group | Intranasal Sufentanil, Pain Relief
Number analyzed (Participants) | 15
Units on a scale | 4.3 (2.2)

ADVERSE EVENTS:
Arm/Group | Intranasal Sufentanil, Pain Relief
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Sufentanil, Pain Relief (N=16)
transient hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — One patient experienced transient, mild hypoxia that resolved with low flow (2 L NC) oxygen after about 20 minutes

LIMITATIONS AND CAVEATS:
A single episode of transient, mild hypoxia that resolved with 2 L nasal canula oxygen and that completely resolved after 20 minutes and no longer required oxygen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes